CLINICAL TRIAL: NCT04391270
Title: A Blended Intervention to Promote Physical Activity, Health and Work Productivity Among Office Employees Using Intervention Mapping: A Study Protocol for a Randomized Controlled Trial
Brief Title: A Blended Intervention to Promote Physical Activity, Health and Work Productivity Among Office Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Gao Yang, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12609919
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Physically Well But Worried
Keywords: physical activity; health promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- web-based intervention group (Experimental): Except "Library", the participants in this group will also have access to the "Intervention" sub-section of the website. It will consist of six sessions delivered every two weeks following the same time schedule as the essay delivery in "Library".
  Interventions: Behavioral: web-based intervention
- blended intervention group (Experimental): Except visiting "Library" and "Intervention" of the website, the participants in this group will also receive three face-to-face workshops (40 min per session) held at their workplaces.
  Interventions: Behavioral: blended intervention
- Control group (No Intervention): The participants in the control group will have access to the "Library" sub-section of the website. General information of MVPA, health and work productivity will be provided with 18 short essays, which can be downloaded and printed out. The information will be factual and non-personally tailored.

INTERVENTIONS:
Behavioral: blended intervention — A blended intervention group combining the web-based components with face-to-face workshops and posters
  Arms: blended intervention group
Behavioral: web-based intervention — A web-based intervention only referred to the use of internet without traditional face-to-face workshops and posters
  Arms: web-based intervention group

SUMMARY:
The primary objective of this study is to examine between-group differences in changes of objectively measured MVPA levels (min/week) among a randomly selected sample of office employees who are physically inactive in Hong Kong.

DETAILED DESCRIPTION:
Regular participation in moderate-to-vigorous physical activity (MVPA) is related to decreased risk of morbidity and mortality. Among working populations, lack of MVPA may also be a risk factor for absenteeism and presenteeism. Both traditional workplace-based and web-based interventions have been suggested as being effective in promoting participation MVPA, health-related outcomes, and work-related productivity. However, several challenges limit their application in real world contexts. A 'blended' intervention approach combining the two intervention strategies is proposed to overcome these limitations. The proposed intervention aims to utilize the blended approach to increase participation in MVPA, health-related outcomes, and work productivity among inactive workers.

Methods: The study will comprise of a three group cluster randomized controlled trial (cluster-RCT), comprising a three-month actual intervention and a nine-month behavioral follow-up period. The three groups will be: a web-based intervention group, a blended intervention group combining the web-based components with face-to-face workshops, and a control group. Physically inactive office employees (N = 141) from will be recruited and randomly assigned to the three groups by cluster randomization. The intervention mapping (IM) framework will be used for selecting and applying effective health behavioural theories and behavioural change techniques (BCTs) to the development, implementation and assessment of the intervention, which will be personally tailored. The primary outcome variable will be objectively measured MVPA using an accelerometer. Secondary outcomes will consist of indices of health including adiposity, blood pressure, blood sugar, blood lipids, self-reported depression, anxiety, stress, and health-related quality of life, and work-related variables including absenteeism and presenteeism.

ELIGIBILITY:
Inclusion Criteria:

* physically inactive (do NOT meet the WHO's recommended MVPA levels)
* office employees in Hong Kong.

Exclusion Criteria:

* participants are engaging other ongoing programs involving MVPA promotion
* if they report any conditions preventing them from being active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
moderate-to-vigorous physical activity (MVPA) levels | baseline, 13 weeks, 25 weeks
  examine between-group differences in changes of objectively measured MVPA levels (min/week) among a randomly selected sample of office employees who are physically inactive in Hong Kong

SECONDARY OUTCOMES:
changes of self-report MVPA levels (min/week) | baseline, 13 weeks, 25 weeks
  To examine between-group differences in changes of self-reported MVPA levels (min/week) in different domains among the sample.
Height in meters | baseline, 13 weeks, 25 weeks
  Height will be measured to the nearest 0.1 cm using a stadiometer.
Weight in kilograms | baseline, 13 weeks, 25 weeks
  Weight will be measured to the nearest 0.1 kg on a calibrated digital balance scale (Seca, max. 200 kg, Germany) with the participants wearing lightweight clothing and no shoes.
Body mass index (BMI, kg/m2) | baseline, 13 weeks, 25 weeks
  Body mass index (BMI, kg/m2) will be calculated from weight and height.
Waist circumference (cm) | baseline, 13 weeks, 25 weeks
  Waist circumference (cm) will be measured midway between the lowest rib margin and the top of the iliac crest at the end of gentle expiration
%Body fat | baseline, 13 weeks, 25 weeks
  %BF will be assessed by a Tanita TBF-410 Body Composition Analyzer (Tanita Corporation, Tokyo, Japan) using foot-to-foot bioelectrical impedance analysis (BIA).
Blood pressure (mmHg) | baseline, 13 weeks, 25 weeks
  Blood pressure will be measured using the Omron M6 Compact (HEM-7000-E, Omron Healthcare Corporation, Kyoto, Japan) following standard measurement protocols.
Hemoglobin A1C (%) | baseline, 13 weeks, 25 weeks
  Hemoglobin A1C will be measured using the Reflotron ® Plus system (Roche Diagnostics, F. Hoffmann-La Roche Ltd., Burgess Hill, UK).
Depression, anxiety and stress | baseline, 13 weeks, 25 weeks
  Depression, anxiety and stress will be measured using the Chinese version of the Depression Anxiety Stress Scale (DASS-21)
Presenteeism | baseline, 13 weeks, 25 weeks
  It will be assessed using presenteeism questions derived from the WHO's Heath and Work Performance Questionnaire (HPO).
High-density lipoprotein (mmol/L) | baseline, 13 weeks, 25 weeks
  high-density lipoprotein will be measured using the Reflotron ® Plus system (Roche Diagnostics, F. Hoffmann-La Roche Ltd., Burgess Hill, UK).
Triglyceride (mmol/L) | baseline, 13 weeks, 25 weeks
  Triglyceride will be measured using the Reflotron ® Plus system (Roche Diagnostics, F. Hoffmann-La Roche Ltd., Burgess Hill, UK).

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Hagger, Dr., Principal Investigator — University of California, Merced; Xiangyan Chen, Dr., Principal Investigator — The Hong Kong Polytechnic University; Xiu Ming Fong, Dr., Principal Investigator — Hong Kong Nang Yan College of Higher Education, Hong Kong, China; Chunqing Zhang, Dr., Principal Investigator — Hong Kong Baptist University
Locations (1):
- Department of Sport, Physical Education, and Health, Kowloon Tong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Wang A, Yu S, Hagger MS, Chen X, Fong SSM, Zhang C, Huang WY, Baker JS, Dutheil F, Gao Y. A blended intervention to promote physical activity, health and work productivity among office employees using intervention mapping: a study protocol for a cluster-randomized controlled trial. BMC Public Health. 2020 Jun 25;20(1):994. doi: 10.1186/s12889-020-09128-z. PMID 32586293

DOCUMENTS (1):
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04391270/ICF_001.pdf